CLINICAL TRIAL: NCT05368467
Title: National Registry and Cohort Study of Pulmonary Vascular Disease
Acronym: NCPVD
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Vice President of Nanjing First Hospital, Director of Cardiovascular Department, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: NMU20220505
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Disease Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: All consecutive consenting patients diagnosed with PH according to specific hemodynamic criteria at participating institutions.
  Interventions: Combination Product: The clinical course and disease management

INTERVENTIONS:
Combination Product: The clinical course and disease management — The clinical course and disease management of pulmonary hypertension patients

SUMMARY:
This is a observational、multicenter, prospective cohort study for patients with pulmonary hypertension (PH). The purposes of this study were to evaluate the etiology、clinical characteristics、treatment modalities, and outcomes of patients with PH；also to set up registration system of PH in China, to build a database of Chinese PH, to establish a web-based international standard data acquisition system for PH and a multicenter clinical research platform. The results of the study will provide a basis for the future national health policy for prevention and treatment of PH.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or previously diagnosed patients with PH.
* Documentation of mean pulmonary arterial pressure (mPAP) >20 mm Hg by right heart catheterization, performed at any time prior to study enrollment.

Exclusion Criteria:

* Have not had documentation of hemodynamic criteria for PH by right heart catheterization at some time preceding study entry and following development of symptoms associated with PH.
* Do not meet the required hemodynamic criteria for entry into the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Pulmonary Hypertension from China based PH centers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
All-cause Death | 5 years

SECONDARY OUTCOMES:
Number of Participants with Clinical Worsening | 5 years
  Clinical worsening during follow-up was defined as worsening PAH or atrial septostomy or listing for lung transplantation or all-cause death. Worsening PAH required the presence of worsening PAH symptoms and a decrease in 6-minute walk distance greater than 15% from baseline and the requirement for additional PAH treatments (all three conditions had to be present).

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Nanjing First Hospital, Nanjing, Jiangsu
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Beijing Anzhen Hospital of Capital Medical University, Beijing
  - China-japan Friendship Hospital, Beijing
  - Xiangya Second Hospital, Central South University, Changsha
  - West China Hospital, Sichuan University, Chendu
  - Nanjing Drum Tower Hospital, Nanjing
  - General Hospital of Northen Theater of Command, Shenyang
  - Tongji Hospital, Huazhong University of Science and Technology, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - First Affiliated Hospital of Xi'An Jiaotong University, Xi'an
  - First Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided